CLINICAL TRIAL: NCT06903091
Title: Efficacy of Automated Text-messaging on Activity Limitation in Participants With Chronic Low Back Pain: a Randomized Controlled Trial
Brief Title: Efficacy of Text-messaging on Activity Limitation in People With Chronic Low Back
Acronym: LOMBATEXT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP241558
Record Dates: First submitted 2025-03-14; First posted 2025-03-30 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Chronic Non-specific Low Back Pain
Keywords: Chronic low back pain; SMS; adherence; therapeutic exercises

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: statisticians will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A : SMS (Experimental): * Face-to-face multidisciplinary rehabilitation sessions,
  * Face-to-face medical and physiotherapy clinical consultation at M3
  * Follow-up:
  * Messages type A (received weekly for the first two weeks, then every 15 days): evaluation of self-program exercise practice and encouragement or reminder of the importance of exercise in the treatment of chronic low-back pain.
  * Messages type B (received monthly): evaluation of APE practice over the past week: "how many times did you do your exercise program last week?". Depending on the response: <3 or ≥ 3 times: participants will receive messages of encouragement or will be asked about the main obstacle encountered (key word); levers adapted to the obstacle will be delivered to them.
  Interventions: Procedure: SMS
- ARM B : Usual follow-up (Active Comparator): * Face-to-face multidisciplinary rehabilitation sessions,
  * Face-to-face medical and physiotherapy clinical consultation at M3.
  Interventions: Procedure: SMS

INTERVENTIONS:
Procedure: SMS — Usual follow-up

SUMMARY:
The main aim of this study was to evaluate the medium-term efficacy of an intervention involving personalized, automated text messaging (SMS), following face-to-face rehabilitation sessions, on activity limitation in people with chronic low back pain. We hypothesize that personalized SMS follow-up, following face-to-face rehabilitation sessions, could reduce activity limitation in people with chronic low back pain. Prospective multicenter randomized controlled trial.

Participants in both groups, experimental and comparator will have 4 face-to-face multidisciplinary rehabilitation sessions.

Participants in the 2 groups will have a face-to-face medical-kinesthetic clinical consultation at M3.

Participants in the experimental group will be monitored by personalized SMS messages over 6 months.

DETAILED DESCRIPTION:
Non-specific low-back pain is one of the leading causes of activity limitation worldwide. Physical exercise is the treatment that has the best proven its efficacy on pain and activity limitation. Adherence to treatment is an essential factor in its effectiveness. Adherence decreases over time and is low in the medium and long term. Lack of patient follow-up is incriminated in poor adherence. Improving the follow-up of chronic low back pain patients appears to be an important lever for improving their function in the medium and long term.

The Memoquest digital solution (Calmedica) solution is based on a conversational robot that generates SMS messages. It integrates an alert and relay system by the therapist.

Participants will be recruited from patients seen in consultation in the physical medicine and rehabilitation (PMR) departments and in the networks of physicians and town-based MKs at the three centers. Randomization will be centralized.

Patients in the 2 groups will have 4 face-to-face multidisciplinary rehabilitation sessions, lasting 1h30 each, over approximately 15 days (2/week over 2 weeks). During these sessions, participants will learn a personalized exercise self-program (APE).

Participants in the 2 groups will have a face-to-face medico-kinesitherapy clinical consultation at M3: the doctor will question the patient about the evolution of his pain, check for the absence of warning signs and assess the tolerance and efficacy of pharmacological treatments, where appropriate. The physiotherapist will question the patient on the completion of the exercises in the self-program, and will provide additional information if necessary. The physiotherapist may also suggest modifications to the exercises to support the participant's progress.

Participants in the experimental group will be monitored by personalized SMS messages, over 6 months: from the end of the face-to-face rehabilitation sessions, they will receive 2 types of messages on their cell phones:

* Messages type A (received weekly for the first two weeks, then every 15 days): exercise reminders and encouragement
* Messages type B (received monthly): assessment of APE practice over the past week: "how many times did you do your exercise program last week?". Depending on the response: <3 or ≥ 3 times: participants will receive messages of encouragement or will be asked about the main obstacle encountered (keyword); levers adapted to the obstacle will be delivered to them. If participants wish to receive further information, they will be directed by a link to the Cochin PRM department website.

If the patient raises the same obstacle during 2 successive exchanges, or if the patient does not respond to the reminder message (48 hours after the initial message), or if the response is not appropriate, the participant will be called on the telephone by an MK taking part in the study.

The participant may withdraw from the study at any time by mentioning

ELIGIBILITY:
Inclusion Criteria:

* People with chronic low back pain (common low back pain, duration of low back pain > 3 months)
* People who own a cell phone and have mastered the basics of using it (consulting and sending sms).
* Person with a moderate to high self-efficacy for exercise score (SEE score ≥ 31/90).
* Patient having signed the study participation consent form. Patient affiliated to a social security scheme or entitled beneficiary

Exclusion Criteria:

* Any other pathology affecting postural stability or voluntary active mobility
* Contraindication to exercise
* Lumbar spine surgery in the 12 months prior to inclusion in the study
* Inability to write, speak or read French
* Psychiatric and/or behavioral disorders
* Current pregnancy (declarative) No inclusion of persons covered by articles L. 1121-5 to L. 1121-8 and L. 1122-1-2 of the French Public Health Code (e.g. minors, protected adults, etc.).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Activity limitation | Month 6 (M6)
  Change in score on the Roland Morris Disability questionnaire (RMDQ, 0 no activity limitation; 24, maximum limitation)

SECONDARY OUTCOMES:
Activity limitation | M3
  Change in RMDQ score
Physical activity | M3 and M6
  Change in overall physical activity measured by pedometer: measurement of average daily activity in the 7 days preceding assessments
Pain intensity | M3 and M6
  Change in pain score measured by numerical scale (at the end of face-to-face supervised PEC
Quality of life | M6
  Change in quality of life measured by the Medical Outcome Study Short Form-12
Adherence | M3 and M6
  Change in adherence score: Exercise Adherence Rating Scale (EARS)
Exercice burden | M3 and M6
  Change in exercise burden score : Exercice Therapy Burden questionnaire (ETBQ)
Self-efficacy | M3 and M6
  Change in self-efficacy for exercise
Level of physical activity (IPAQ) | D0 and M6
Perception of change | M6

CONTACTS AND LOCATIONS:
Overall Officials: Camille Camille, MK, Principal Investigator — Université Paris Cité, Faculté de Santé | UFR de Médecine
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Service de Rééducation et de Réadaptation de l'Appareil Locomoteur et des Pathologies du Rachis, Hôpital Cochin, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No